CLINICAL TRIAL: NCT01181167
Title: A Phase 3, Randomized, Double-Blind, Double-Dummy Efficacy and Safety Study of the Oral Factor Xa Inhibitor DU-176b Compared With Enoxaparin Sodium for Prevention of Venous Thromboembolism in Patients After Total Hip Arthroplasty (STARS J-5 Trial)
Brief Title: A Study of DU-176b, Prevention of Venous Thromboembolism in Patients After Total Hip Arthroplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DU176b-B-J304
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2015-02

CONDITIONS: Prevention; Venous Thromboembolism
Keywords: Anticoagulants; Venous thromboembolism; Thromboembolism; Thrombosis; enoxaparin sodium; Embolism; Deep vein thrombosis; DU-176b; edoxaban; factor Xa; total hip arthroplasty
MeSH Terms: conditions — Venous Thromboembolism; Thromboembolism; Thrombosis; Embolism; Venous Thrombosis | interventions — edoxaban; enoxaparin sodium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- DU-176b (Experimental): DU-176b oral tablets, 30 mg., taken once daily for 2 weeks, initiated within 6 to 24 hours after surgery.
  Interventions: Drug: edoxaban
- enoxaparin sodium (Active Comparator): enoxaparin sodium 20mg(=2000IU)/0.2ml twice daily, subcutaneous injection for 2 weeks, initiated within 24 to 36 hours after surgery.
  Interventions: Drug: enoxaparin sodium

INTERVENTIONS:
Drug: edoxaban
  Arms: DU-176b
Drug: enoxaparin sodium
  Arms: enoxaparin sodium

SUMMARY:
The objective of this study is to assess the efficacy and safety of DU-176b compared with enoxaparin sodium for the prevention of venous thromboembolism in patients after elective total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral total hip arthroplasty

Exclusion Criteria:

* Subjects with risks of hemorrhage
* Subjects with thromboembolic risks
* Subjects who weigh less than 40 kg
* Subjects who are pregnant or suspect pregnancy, or subjects who want to become pregnant

Ages: 20 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Actual)
Dates: Start 2009-05; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Fuji, Principal Investigator — Osaka Koseinenkin Hospital
Locations (2):
- Japan (2):
  - Osaka
  - Tokyo

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Kawai Y, Fuji T, Fujita S, Kimura T, Ibusuki K, Abe K, Tachibana S. Edoxaban versus enoxaparin for the prevention of venous thromboembolism after total knee or hip arthroplasty: pooled analysis of coagulation biomarkers and primary efficacy and safety endpoints from two phase 3 trials. Thromb J. 2016 Dec 1;14:48. doi: 10.1186/s12959-016-0121-1. eCollection 2016. PMID 27980462

RESULTS

PARTICIPANT FLOW:
Groups:
- DU-176b: DU-176b oral tablets, 30 mg., taken once daily for 2 weeks
  edoxaban
- Enoxaparin Sodium: enoxaparin sodium 20mg(=2000IU)/0.2ml twice daily, subcutaneous injection for 2 weeks
  enoxaparin sodium
Period: Overall Study
Arm/Group | DU-176b | Enoxaparin Sodium
Started | 307 | 303
Efficacy Analysis Population | 255 | 248
Completed | 284 | 271
Not Completed | 23 | 32
Not completed — Adverse Event | 11 | 21
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 2 | 3
Not completed — Protocol Violation | 3 | 0
Not completed — Withdrawal by Subject | 6 | 8

BASELINE CHARACTERISTICS:
Population: Number of baseline participants reflects the efficacy analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | DU-176b | Enoxaparin Sodium | Total
Number analyzed (Participants) | 255 | 248 | 503
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (9.61) | 62.8 (9.72) | 62.8 (9.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 220 | 212 | 432
  Male | 35 | 36 | 71
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 255 | 248 | 503
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 255 | 248 | 503

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Subjects With Venous Thromboembolism Events
Description: The primary efficacy endpoint was the proportion of subjects who experienced at least one of the thromboembolic events listed below during the period from the start of study treatment to the venography at the end of study treatment.
  * Lower extremity DVT confirmed by bilateral venography at the end of study treatment
  * Definite diagnosis of symptomatic PE
  * Symptomatic DVT confirmed before the venography at the end of study treatment The objectives were to verify the non-inferiority of edoxaban to enoxaparin with regard to prevention of VTE
Time Frame: 2 weeks
Population: The FAS was defined as all subjects enrolled in the study, but excluded those who had significant GCP violations, who had not received any doses of the study drug, or those who did not develop symptomatic DVT or PE, but in whom venography was not appropriately performed.
Measure: Number (95% Confidence Interval); unit: percentage of subjects with vte events
Arm/Group | DU-176b | Enoxaparin Sodium
Number analyzed (Participants) | 255 | 248
percentage of subjects with vte events | 2.4 [1.1 to 5.0] | 6.9 [4.3 to 10.7]
Statistical Analysis 1: Comparison: DU-176b vs Enoxaparin Sodium; Hypothesis testing of proportion of subjects who experienced at least one thromboembolic events, defined as primary endpoint, carried out using Farrington-Manning method. Null hypothesis H˅01: Incidence of thromboembolic events in DU-176b group (P˅DU) = Incidence of thromboembolic events in enoxaparin group (P˅E) + Δ (8%). Alternative hypothesis H˅11: P˅DU < P˅E + Δ (significance level: One-sided, 0.025); Test type: Non-Inferiority or Equivalence — Difference in incidence of thromboembolic events between DU-176b and enoxaparin groups and 95% confidence interval (CI) were calculated. Incidence of thromboembolic events and 95% CI also calculated by treatment group. Only when null hypothesis H01 was rejected, upper limit of 95% CI for difference between DU-176b and enoxaparin groups was confirmed. When upper limit of 95% CI was below 0%, DU-176b was considered to be superior to enoxaparin in terms of the prevention of VTE; p < 0.001, ANCOVA — Farrington Manning Method; Cox Proportional Hazard = -4.5

2. Secondary Outcome: Incidence of Major Bleeding or Clinically Relevant Non-major Bleeding
Time Frame: 2 weeks
Population: Safety analyses were performed for the Safety Analysis Set, which was defined as all subjects who were secondarily enrolled in the study, but excluded those who had significant GCP violations, who had not received any doses of the study drug, or who had no safety data after the start of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of subjects with bleeds
Arm/Group | DU-176b | Enoxaparin Sodium
Number analyzed (Participants) | 303 | 301
percentage of subjects with bleeds | 2.6 [1.3 to 5.1] | 3.7 [2.1 to 6.7]

ADVERSE EVENTS:
Arm/Group | DU-176b | Enoxaparin Sodium
Serious Adverse Events (participants affected / at risk) | 9/303 | 9/301
Other Adverse Events (participants affected / at risk) | 197/303 | 232/301
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DU-176b (N=303) | Enoxaparin Sodium (N=301)
deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
otrhostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0)
intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
abcess jaw (Infections and infestations) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DU-176b (N=303) | Enoxaparin Sodium (N=301)
Aspartate aminotransferase increased (Investigations) | 17 (17) | 97 (98)
Gamma-glutamyltransferase increased (Investigations) | 44 (45) | 79 (81)
Alanine aminotransferase increased (Investigations) | 36 (37) | 126 (128)
Blood urine present (Investigations) | 38 (39) | 34 (37)
Blood alkaline phosphatase increased (Investigations) | 14 (15) | 40 (41)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 12 (12) | 21 (23)
Blood bilirubin increased (Investigations) | 11 (11) | 10 (10)
headache (Nervous system disorders) | 11 (12) | 12 (12)
Abdominal discomfort (Gastrointestinal disorders) | 9 (10) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 10 (10) | 10 (10)
Haematuria (Renal and urinary disorders) | 11 (12) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall not publish the results of the Study at any time without the prior written approval of Sponsor.